CLINICAL TRIAL: NCT05526833
Title: An Open-label Extension Trial of Individualized Repetitive Transcranial Magnetic Stimulation in Patients With Auditory Verbal Hallucinations Who Completed Protocol #8116
Brief Title: An Extension Protocol for Patients Who Previously Completed the TMS Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator departed from institution
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8249; K23MH119318 (NIH)
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia and Related Disorders
Keywords: Hallucinations; Auditory Verbal Hallucinations
MeSH Terms: conditions — Schizophrenia; Hallucinations | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Schizophrenia patients with AVH who have completed protocol #8116 will be recruited, and allocated to one of three arms based on their treatment responsiveness from protocol #8116 which included 10 low-frequency TMS treatment sessions using the TPJ target. Their treatment responsiveness is assessed by the Auditory Hallucination Rating Scale (AHRS) at pre- and post-TMS session. Non-responders will be offered 10 daily sessions of 1-Hz rTMS delivered to the rSTS region instead. Partial responders will be offered 10 additional daily sessions of 1-Hz rTMS delivered to the same original left TPJ target used in protocol #8116. Full responders will be offered followup clinical assessments at 1,2,4, and 8 weeks to assess sustainability of their response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Non-responders undergo rTMS of the right superior temporal sulcus (STS) (Experimental): Non-responders to protocol #8116 will receive a type of TMS called repetitive TMS (rTMS) wherein the magnetic pulses delivered will be close together in a rapid sequence. They will be administered 10 days (10 sessions) of MRI-guided 1 Hz rTMS delivered to the right superior temporal sulcus (STS). The rTMS parameters that will be used are a frequency of 1 Hz (1 pulse per second) at an intensity of 90% of the motor threshold (MT). Therefore, the investigators will deliver 1200 continuous pulses per session/day which adds up to 12,000 pulses in total for the whole treatment.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Partial responders undergo rTMS of the left temporo-parietal junction (TPJ) (Experimental): Partial responders to protocol #8116 will receive a type of TMS called repetitive TMS (rTMS) wherein the magnetic pulses delivered will be close together in a rapid sequence. They will be administered 10 days (10 sessions) of MRI-guided 1 Hz rTMS delivered to the original left temporo-parietal junction (TPJ) target. The rTMS parameters that will be used are a frequency of 1 Hz (1 pulse per second) at an intensity of 90% of the motor threshold (MT). Therefore, the investigators will deliver 1200 continuous pulses per session/day which adds up to 12,000 pulses in total for the whole treatment.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Complete responders undergo four follow-up clinical assessments (No Intervention): Complete responders to protocol #8116 will be offered followup clinical assessments at 1, 2, 4, and 8 weeks to assess sustainability of their response.

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — During the rTMS session, an electromagnetic coil is placed on the scalp of the subject's head. The electromagnet painlessly delivers a magnetic pulse that stimulates nerve cells in the region of the brain involved in speech perception.
  Arms: Non-responders undergo rTMS of the right superior temporal sulcus (STS); Partial responders undergo rTMS of the left temporo-parietal junction (TPJ)

SUMMARY:
This is an open-label extension study to continue to evaluate the safety, tolerability and efficacy of the Repetitive Transcranial Magnetic Stimulation (rTMS) in subjects with schizophrenia or schizoaffective disorder who previously completed the treatment study of the protocol #8116 (NCT05319080). Protocol #8116 investigates the clinical efficacy of open-label individualized MRI-guided TMS applied to the left temporoparietal junction (TPJ) in schizophrenia patients. Participating patients who have completed the 4-week project #8116 can be screened for eligibility for this extension study in which they will continue treatment/assessment. They will be divided into three groups (non-responders, partial responders, or full responders) based on a reduction in the Auditory Hallucination Rating Scale (AHRS) scores from the study #8116.

DETAILED DESCRIPTION:
The optimal neuroanatomical treatment targets remain unclear, though current neuroscience evidence suggests several brain areas such as the left temporo-parietal junction area (TPJ) or the right posterior superior temporal sulcus (rSTS) may be involved in the generation and development of AVH. During this extension study, non-responders to protocol #8116 will be administered 10 days (10 sessions) of MRI-guided 1 Hz rTMS delivered to the rSTS instead of the original target in TPJ. Partial responders will receive 10 additional low-frequency rTMS over the original left TPJ target. Like the protocol #8116, the investigators will use the MRI-guided targeting approach during rTMS treatment sessions to achieve greater precision as it can account for individual differences in anatomy. Complete responders will instead be followed for sustainability of response. Their clinical ratings will be repeated at one week, two week, four week and eight week follow-ups. Non-responders are defined as patients showing a reduction of AHRS less than 20% of the initial score. A partial response is defined as a reduction in a range of between 20% and 50% of the initial AHRS score. A complete response is defined as a reduction by at least 50% of the initial AHRS score.The combined outcome of protocol #8116 and the currently proposed protocol will help guide TMS targeting and the number of treatment sessions for a future larger randomized, double-blinded, shame-controlled clinical trial.

ELIGIBILITY:
For non responders and partial responders:

Inclusion Criteria:

* Completion of the study #8116 (NCT05319080)
* The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of schizophrenia or schizoaffective disorder
* A reduction of AHRS less than 50% of the initial score
* Capacity and willingness to provide informed consent
* If female and not infertile, must agree to use one of the following forms of contraception for the duration of study participation: systemic hormonal treatment, an intrauterine device (IUD) which was implanted at least 2 months prior to screening, or "double-barrier" contraception. Women of child bearing potential must have a negative pregnancy test at screening
* Right handed
* Normal hearing
* Taking an antipsychotic medication at a stable dose for at least 4 weeks. All oral and depot antipsychotics are allowable.

Exclusion Criteria:

* Substance use disorder (excluding nicotine) within last 90 days, or positive toxicology screen for any substance of abuse
* Pregnancy
* Severe adverse events of TMS
* History of seizure, epilepsy and neurologic conditions with structural cerebral damage, including stroke, multiple sclerosis, traumatic brain injury, Alzheimer's and other neurodegenerative diseases, meningoencephalitis or intracerebral abscess, parenchymal or leptomeningeal cancers, dementia, developmental disability, cerebrovascular disease, increased intracranial pressure, or central nervous system (CNS) tumors, brain surgery, head injury with loss of consciousness >1 hour or clear cognitive sequelae, intracranial metal implants, known structural brain lesion
* Subjects with devices that may be affected by TMS (pacemaker, cardioverter defibrillator, medication pump, intracardiac line, cochlear implant, implanted brain stimulator/neurostimulator)
* Subjects with suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the Suicidal Ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the investigator
* Frequent and persistent migraines
* Clinically significant skin disease
* Presence of unstable medical disorders, including those that are previously undiagnosed, untreated, inadequately treated, or active to an extent which might make participation hazardous. For example, hypertension, previous stroke, brain lesions, or heart disease
* History of prior clinically significant, adverse response to neurostimulation
* Current treatment with ototoxic medications (amino-glycosides, cisplatin)

For complete responders:

Inclusion Criteria:

* Completion of the study #8116 (NCT05319080)
* The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of schizophrenia or schizoaffective disorder
* A reduction by at least 50% of the initial AHRS score
* Taking an antipsychotic medication at a stable dose for at least 4 weeks. All oral and depot antipsychotics are allowable.

Exclusion Criteria:

* Substance use disorder (excluding nicotine) within last 90 days, or positive toxicology screen for any substance of abuse
* Subjects with suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the Suicidal Ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the investigator
* Presence or positive history of unstable significant medical or neurological illness

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Avissar, MD, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Started | 1 | 1 | 1
Completed | 1 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants] — Population: As N=1 for each arm, the baseline charactertistics are not being disclosed to protect the confidentiality of the participants.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: As N=1 for each arm, the baseline charactertistics are not being disclosed to protect the confidentiality of the participants.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: As N=1 for each arm, the baseline charactertistics are not being disclosed to protect the confidentiality of the participants.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Number of rTMS Sessions Completed
Description: The total number of rTMS sessions completed for non responders and partial responders. A session is defined as 20 minutes of rTMS.
Time Frame: 2 weeks.
Population: Zero participants analyzed as n=1 for each arm. Results are not included here to protect the confidentiality of the participants.
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Total Number of Follow-up Clinical Assessments Completed
Description: The total number of follow-up clinical assessments completed for complete responders. A clinical assessment refers to answering questions about psychiatric symptoms to assess the sustainability of the patient's improvement from the previous study.
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Total Number of Treatment Emergent Adverse Events
Description: The total number of treatment emergent adverse events for non responders and partial responders. An emergent adverse event is defined as any rTMS risk induced incident in research such as headache and seizure.
Time Frame: 2 weeks.
Population: as for outcome 1
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in Auditory Hallucination Rating Scale (AHRS)
Description: The AHRS is an investigator-administered scale assessing multiple characteristics of auditory verbal hallucinations. The total score ranges from 2 to 41, with higher scores indicating more severe symptoms.
Time Frame: Up to 4/8 weeks.
Population: as for outcome 1
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change in Psychotic Symptom Rating Scale (PSYRATS)
Description: The PSYRATS consists of 17 items on delusions and auditory hallucinations, with each item being rated from 0 (absent) to 4 (severe). The total score ranges from 0 to 68, with higher scores indicating more severe symptoms.
Time Frame: Up to 4/8 weeks.
Population: as for outcome 1
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change in Scale for the Assessment of Positive Symptoms (SAPS)
Description: The SAPS includes 34 items that focus on the positive symptoms on schizophrenia. Each item is rated from o to 5 (range=0-170). Higher scores indicate more severe symptoms.
Time Frame: Up to 4/8 weeks.
Population: as for outcome 1
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS)
Description: The PANSS rates the presence and severity of positive and negative symptoms, as well as general psychopathology associated with schizophrenia. Each item is rated from 1 to 7 (range=30-210). Higher scores indicate more severe symptoms.
Time Frame: Up to 4/8 weeks.
Population: as for outcome 1
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change in Cardiff Anomalous Perceptions Scale (CAPS)
Description: The CAPS is a 32 item scale for measuring perceptual anomalies, that includes subscales for measuring distress, intrusiveness and frequency. A higher score indicates a higher number of perceptual anomalies, scores range from 0 (low) to 32 (high).
Time Frame: Up to 4/8 weeks.
Population: as for outcome 1
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change in Clinical Global Impression Improvement (CGI-I) Scale
Description: The CGI-I is a clinician-rated scale to quantify overall clinician impression of improvements in level of illness. The CGI-I is rated on a 7-point scale, to assess illness improvement. CGI-I scores range from 1 (very much improved) through to 7 (very much worse).
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Change in Clinical Global Impression Severity (CGI-S) Scale
Description: The CGI-S is a clinician-rated scale to quantify overall clinician impression of illness severity. The CGI-S is rated on a 7-point scale, to assess illness severity. CGI-S scores range from 1 (normal, not ill) through to 7 (among the most severely ill patients).
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: As n=1 per arm, data is not disclosed to protect participant confidentiality.
Arm/Group | Non-responders Undergo rTMS of the Right Superior Temporal Sulcus (STS) | Partial Responders Undergo rTMS of the Left Temporo-parietal Junction (TPJ) | Complete Responders Undergo Four Follow-up Clinical Assessments
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study ended prematurely, resulting in a sample size that did not meet our expectations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT05526833/Prot_002.pdf
  • Informed Consent Form (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT05526833/ICF_001.pdf